CLINICAL TRIAL: NCT03682913
Title: Personalized Inhibitory Control Training for Compulsive Behavior Change
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hebrew University of Jerusalem (Other)
Responsible Party: Principal Investigator, Shahaf Leshem, Principal investigator, Hebrew University of Jerusalem
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0105-18-HMO
Record Dates: First submitted 2018-08-23; First posted 2018-09-25 (Actual); Last update posted 2018-09-27 (Actual); Status verified 2018-09

CONDITIONS: OCD

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- P-CIT protocol (Experimental): OCD patients who receive the P-CIT intervention.
  Interventions: Behavioral: P-CIT protocol
- Placebo (Placebo Comparator): OCD patients who don't receive the P-CIT intervention.
  Interventions: Behavioral: Placebo

INTERVENTIONS:
Behavioral: P-CIT protocol — Personalized inhibitory control training for one week.
  Arms: P-CIT protocol
Behavioral: Placebo — without personalized inhibitory control training for one week.
  Arms: Placebo

SUMMARY:
Obsessive-compulsive disorder (OCD) is a severe mental illness characterized by repetitive behaviors that a person feels compelled to perform. It has been demonstrated that stimuli in the environment can trigger the compulsive urge, perpetuating the OCD cycle. The main goal of the current proposal, which is based on exciting pilot data, is to test a novel computerized training program to create an association between OCD-related stimuli, which typically trigger the compulsive urge, and the brain system responsible for stopping. The idea is that once this system is triggered, it will be easier for patients to stop the compulsive urge.

ELIGIBILITY:
Inclusion Criteria:

* OCD patients

Exclusion Criteria:

* Metal/ electronic device
* Under the age of 18
* Pregnant women
* Tattoos that cover over 10% of body mass
* Chronically ill patients
* Psychosis/ Bi-polar
* Substance abuse
* Sever depression
* Active suicide thoughts
* Hearing loss

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-07-30 (Estimated); Study Completion 2019-08-30 (Estimated)

PRIMARY OUTCOMES:
fMRI- changed inhibition levels in the pre-SMA area in experimental group in comparison to control group | One week after P-CIT training starts
  During tasks that require inhibition
fMRI- changed inhibition levels in the rIFG area in experimental group in comparison to control group | One week after P-CIT training starts
  During tasks that require inhibition

SECONDARY OUTCOMES:
Behavioural- Y-bocs (Yale-Brown Obsessive-Compulsive Scale) score- change in OCD symptoms in experimental group in comparison to placebo group | One week after P-CIT (Personalized Inhibitory Control Training for Compulsive Behavior Change) training
  Clinical assessment. Semi-structured interview that assesses the presence and severity of obsessions and compulsions over the past week. The 5-item Obsession Severity and Compulsion Severity subscales are summed to produce a Total Severity score. Symptoms endorsed are rated on a scale from none (0) to extreme (5). The 5-item Obsession Severity and Compulsion Severity subscales are summed to produce a Total Severity score.
Behavioural- M.I.N.I (Mini-International Neuropsychiatric Interview) score- change in OCD symptoms in experimental group in comparison to placebo group | One week after P-CIT (Personalized Inhibitory Control Training for Compulsive Behavior Change) training
  Clinical assessment. Structural interview.
Behavioural- OCI-R (Obsessive-Compulsive Inventory) score- change in OCD symptoms in experimental group in comparison to placebo group | One week after P-CIT (Personalized Inhibitory Control Training for Compulsive Behavior Change) training
  Clinical assessment. Cutoff score of 21 is distinguish individuals with OCD from those without anxiety disorders.

CONTACTS AND LOCATIONS:
Locations (1):
- The Hebrew University of Jerusalem, Jerusalem, Israel